CLINICAL TRIAL: NCT00518882
Title: Effect of Liraglutide or Exenatide Added to a Background Treatment of Metformin, Sulphonylurea or a Combination of Both on Glycaemic Control in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide or Exenatide Added to an Ongoing Treatment on Blood Glucose Control in Subjects With Type 2 Diabetes
Acronym: LEAD-6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1797; 2006-006092-21 (EudraCT Number)
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Results first posted 2010-03-23 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide 1.8 mg once daily + subject's own OAD treatment
  Interventions: Drug: liraglutide
- Exenatide (Active Comparator): Exenatide 10 mcg twice daily + subject's own OAD treatment
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: liraglutide — 1.8 mg once daily for s.c. (under the skin) injection.
  Arms: Liraglutide
Drug: exenatide — 10 mcg twice daily for s.c. (under the skin) injection.
  Arms: Exenatide

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to compare the effect on glycaemic control of liraglutide or exenatide when added to subject's ongoing OAD (oral anti-diabetic drug) treatment of either metformin, sulphonylurea or a combination of both in subjects with type 2 diabetes. Two trial periods: A 26 week randomised, followed by a 52 week extension (14 + 38 weeks) where all subjects received liraglutide + OAD after previous randomisation to either liraglutide or exenatide, both combined with OAD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Stable treatment with Oral Anti-Diabetic Drugs (metformin, sulphonylurea or a combination of both) for at least 3 months at the discretion of the Investigator
* HbA1C equal to or greater than 7.0% and equal to or lower than 11.0%
* Body Mass Index (BMI) equal to or lower than 45.0 kg/m2

Exclusion Criteria:

* Previous treatment with insulin
* Treatment with any anti-diabetic drug other than metformin and sulphonylurea
* Any previous exposure to exenatide or liraglutide
* Impaired liver or/and renal function
* History of any significant cardiac events
* Known retinopathy or maculopathy requiring acute treatment
* Recurrent major hypoglycaemia or hypoglycaemic unawareness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (116):
- United States (57):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Artesia, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Fort Myers, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Longwood, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Saint Cloud, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Powder Springs, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Saint Paul, Minnesota
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Flemington, New Jersey
  - Novo Nordisk Investigational Site, South Bound Brook, New Jersey
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Canton, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Sumter, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Vienna
- Denmark (5):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Odense
- Finland (3):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Oulu
- France (5):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Dommartin-lès-Toul
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
- Germany (14):
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Dreieich-Sprendlingen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Herrenberg
  - Novo Nordisk Investigational Site, Lampertheim
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Tübingen
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Norway (3):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Poland (9):
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Gniewkowo
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Tychy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
  - Novo Nordisk Investigational Site, Zabrze
- Novo Nordisk Investigational Site, Manatí, Puerto Rico
- Romania (3):
  - Novo Nordisk Investigational Site, Alba Iulia, Alba
  - Novo Nordisk Investigational Site, Suceava, Suceava
  - Novo Nordisk Investigational Site, Reşiţa
- Slovenia (3):
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Novo Mesto
- Spain (4):
  - Novo Nordisk Investigational Site, L'Hospitalet de Llobregat
  - Novo Nordisk Investigational Site, Oviedo
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Puerto del Rosario
- Novo Nordisk Investigational Site, Stockholm, Sweden
- Switzerland (4):
  - Novo Nordisk Investigational Site, Basel
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lugano

REFERENCES:
- [Result] Sullivan SD, Alfonso-Cristancho R, Conner C, Hammer M, Blonde L. Long-term outcomes in patients with type 2 diabetes receiving glimepiride combined with liraglutide or rosiglitazone. Cardiovasc Diabetol. 2009 Feb 26;8:12. doi: 10.1186/1475-2840-8-12. PMID 19245711
- [Result] McGill JB. Insights from the Liraglutide Clinical Development Program--the Liraglutide Effect and Action in Diabetes (LEAD) studies. Postgrad Med. 2009 May;121(3):16-25. doi: 10.3810/pgm.2009.05.1998. PMID 19491536
- [Result] Buse JB, Rosenstock J, Sesti G, Schmidt WE, Montanya E, Brett JH, Zychma M, Blonde L; LEAD-6 Study Group. Liraglutide once a day versus exenatide twice a day for type 2 diabetes: a 26-week randomised, parallel-group, multinational, open-label trial (LEAD-6). Lancet. 2009 Jul 4;374(9683):39-47. doi: 10.1016/S0140-6736(09)60659-0. Epub 2009 Jun 8. PMID 19515413
- [Result] Buse JB, Sesti G, Schmidt WE, Montanya E, Chang CT, Xu Y, Blonde L, Rosenstock J; Liraglutide Effect Action in Diabetes-6 Study Group. Switching to once-daily liraglutide from twice-daily exenatide further improves glycemic control in patients with type 2 diabetes using oral agents. Diabetes Care. 2010 Jun;33(6):1300-3. doi: 10.2337/dc09-2260. Epub 2010 Mar 23. PMID 20332351
- [Result] Schmidt WE, Christiansen JS, Hammer M, Zychma MJ, Buse JB. Patient-reported outcomes are superior in patients with Type 2 diabetes treated with liraglutide as compared with exenatide, when added to metformin, sulphonylurea or both: results from a randomized, open-label study. Diabet Med. 2011 Jun;28(6):715-23. doi: 10.1111/j.1464-5491.2011.03276.x. PMID 21388442
- [Result] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Result] Valentine WJ, Palmer AJ, Lammert M, Langer J, Brandle M. Evaluating the long-term cost-effectiveness of liraglutide versus exenatide BID in patients with type 2 diabetes who fail to improve with oral antidiabetic agents. Clin Ther. 2011 Nov;33(11):1698-712. doi: 10.1016/j.clinthera.2011.09.022. Epub 2011 Oct 21. PMID 22018679
- [Result] Bode BW, Brett J, Falahati A, Pratley RE. Comparison of the efficacy and tolerability profile of liraglutide, a once-daily human GLP-1 analog, in patients with type 2 diabetes >/=65 and <65 years of age: a pooled analysis from phase III studies. Am J Geriatr Pharmacother. 2011 Dec;9(6):423-33. doi: 10.1016/j.amjopharm.2011.09.007. Epub 2011 Nov 4. PMID 22055210
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Result] Davidson JA, Orsted DD, Campos C. Efficacy and safety of liraglutide, a once-daily human glucagon-like peptide-1 analogue, in Latino/Hispanic patients with type 2 diabetes: post hoc analysis of data from four phase III trials. Diabetes Obes Metab. 2016 Jul;18(7):725-8. doi: 10.1111/dom.12653. Epub 2016 Apr 28. PMID 26936426
- [Derived] Fonseca VA, Devries JH, Henry RR, Donsmark M, Thomsen HF, Plutzky J. Reductions in systolic blood pressure with liraglutide in patients with type 2 diabetes: insights from a patient-level pooled analysis of six randomized clinical trials. J Diabetes Complications. 2014 May-Jun;28(3):399-405. doi: 10.1016/j.jdiacomp.2014.01.009. Epub 2014 Jan 21. PMID 24561125
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 133 centres in 15 countries: Austria (4), Denmark (6), Finland (5), France (5), Germany (14), Ireland (4), Macedonia (1), Norway (4), Poland (9), Romania (3), Slovenia (3), Spain (4), Sweden (2), Switzerland (4) and United States (65).
Pre-assignment Details: Eligible subjects were subjects with type 2 diabetes being treated with oral anti-diabetic (OAD) therapy(ies) for at least 3 months prior to the study. Three subjects were exposed to study drug prior to randomisation, and thus only included in safety analysis set.
Groups:
- Liraglutide -> Liraglutide -> Liraglutide: Liraglutide 1.8 mg once daily + OAD (metformin monotherapy, sulphonylurea (SU) monotherapy or a combination), Weeks 0-26 (double-blinded) continued to receive liraglutide 1.8 mg once daily + OAD in extension period (weeks 26-52 and 52-78)
- Exenatide -> Liraglutide -> Liraglutide: Exenatide 10 mcg twice daily + OAD (metformin monotherapy, sulphonylurea (SU) monotherapy or a combination), Weeks 0-26 (double-blinded) switched to receive liraglutide 1.8 mg once daily + OAD in extension period (weeks 26-52 and 52-78)
Period: Double-Blind, Week 0-26
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Started | 235 (2 subjects exposed to study drug before randomisation. Subjects only included in safety analysis set) | 232 (1 subject exposed to study drug before randomisation. Subject only included in safety analysis set)
Randomised | 233 | 231
Completed | 202 | 187
Not Completed | 33 | 45
Not completed — Adverse Event | 23 | 31
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal criteria | 1 | 1
Not completed — Lost to follow up | 2 | 1
Not completed — Subject decision | 1 | 1
Not completed — Withdrawal of consent | 1 | 3
Not completed — Loss of trust | 0 | 1
Not completed — Fear of hypoglycaemia | 0 | 1
Not completed — Hypoglycaemia | 0 | 2
Not completed — Mutual consent | 0 | 1
Period: Open-Label Extension, Week 26-78
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Started | 202 | 187
Completed | 161 | 138
Not Completed | 41 | 49
Not completed — Adverse Event | 3 | 9
Not completed — Lack of Efficacy | 6 | 5
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawel criteria | 1 | 2
Not completed — Hypoglycaemia | 0 | 1
Not completed — Lost to follow up | 1 | 1
Not completed — Consent withdrawn | 2 | 1
Not completed — Change in treatment | 1 | 1
Not completed — Creatine increased | 1 | 0
Not completed — Decreased kidney function | 1 | 0
Not completed — Exclusion criteria | 2 | 0
Not completed — Subject decision | 2 | 0
Not completed — Completed extension 1 (weeks 26-40) | 18 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide | Total
Number analyzed (Participants) | 233 | 231 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.8) | 57.1 (10.8) | 56.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 104 | 223
  Male | 114 | 127 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 25 | 57
  Not Hispanic or Latino | 201 | 206 | 407
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 12 | 25
  White | 216 | 210 | 426
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Previous OAD treatment [Number; unit: participants] — OAD = Oral Anti-diabetic Drug
  participants
    Metformin/Sulphonylurea Combination | 145 | 147 | 292
    Sulphonylurea | 24 | 21 | 45
    Metformin | 64 | 63 | 127
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 32.9 (5.5) | 32.9 (5.7) | 32.9 (5.6)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 8.5 (6.2) | 7.9 (5.9) | 8.2 (6.0)
HbA1c [Mean (Standard Deviation); unit: percentage of total haemoglobin] — Glycosylated Haemoglobin at screening
  percentage of total haemoglobin | 8.4 (1.0) | 8.2 (1.0) | 8.3 (1.0)
Height [Mean (Standard Deviation); unit: m] | 1.68 (0.10) | 1.68 (0.10) | 1.68 (0.10)
Weight [Mean (Standard Deviation); unit: kg] | 93.1 (20.1) | 93.0 (19.5) | 93.1 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated A1c (HbA1c) at Week 26
Description: Percentage point change in glycosylated A1c (HbA1c) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: Intention to Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects exposed to study drug.
Measure: Least Squares Mean (Standard Error); unit: percentage point of total HbA1c
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 227 | 226
percentage point of total HbA1c | -1.12 (0.08) | -0.79 (0.08)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; ANCOVA with treatment, country and previous OAD treatment as fixed effects and baseline HbA1c as covariate. 2 hypotheses were tested: H01: µliraglutide ≥ µexenatide + Δ, HA1: µliraglutide < µexenatide + Δ; Δ=0.4%. If non-inferiority was concluded, a test for superiority was established by a 1-sided test of the hypothesis H02: µliraglutide ≥ µexenatide against HA2: µliraglutide < µexenatide. Superiority was concluded if the upper limit of the 2-sided 95% CI for the difference was below 0%; Test type: Non-Inferiority or Equivalence — Non-inferiority concluded if upper confidence interval of test is below 0.4%; p < .0001, ANCOVA — No multiplicity concerns; Estimated treatment difference, LS Mean = -0.33, 95% CI [-0.47 to -0.18]

2. Secondary Outcome: Change in Glycosylated A1c (HbA1c), Weeks 26-78
Description: Percentage point change in glycosylated A1c (HbA1c) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group)
Time Frame: week 26, week 78
Population: Intention to Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects who entered the extension period and who had been exposed to at least one dose of the study drugs.
Measure: Mean (Standard Deviation); unit: percentage point of total HbA1c
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 183
percentage point of total HbA1c | 0.25 (0.803) | -0.00 (0.924)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; A paired t test was made within the treatment group and 95% confidence intervals for the difference between Weeks 26 and 78 were constructed. H0 was µ78 - µ26 = 0 against HA: µ78 - µ26 ≠ 0. A difference between the two means (Week 26 and Week 78) was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean = 0.25, 95% CI [0.139 to 0.364], Standard Deviation 0.803
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9872, Paired t-test; Mean = -0.00, 95% CI [-1.36 to 0.134], Standard Deviation 0.924

3. Secondary Outcome: Change in Glycosylated A1c (HbA1c) at Week 78
Description: Percentage point change in glycosylated A1c (HbA1c) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group)
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage point of total HbA1c
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 183
percentage point of total HbA1c | -0.98 (1.119) | -0.85 (1.105)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; The analysis was made with a paired t test within the treatment group and 95% confidence intervals for the difference between Weeks 0 and 78 were constructed. H0 was µ78 - µ0 = 0 against HA: µ78 - µ0 ≠ 0. A difference between the two means (Weeks 0 and 78) was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean = -0.98, 95% CI [-1.137 to -0.823], Standard Deviation 1.119
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; The analysis was made with a paired t test within the exenatide→liraglutide group and 95% confidence intervals for the difference between Weeks 0 and 78 were constructed. H0 was µ78 - µ0 = 0 against HA: µ78 - µ0 ≠ 0. A difference between the two means (Weeks 0 and 78) was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean = -0.85, 95% CI [-1.010 to -0.687], Standard Deviation 1.105

4. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of Either HbA1c < 7.0% or =< 6.5% at Week 26
Description: Percentage of subjects achieving treatment target of HbA1c less than 7.0% or less than or equal to 6.5% at Week 26 (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 233 | 231
percentage (%) of subjects
  Treatment target HbA1c < 7% | 53 | 42
  Treatment target HbA1c =< 6.5% | 34 | 20

5. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of Either HbA1c < 7.0% or =< 6.5% at Week 78
Description: Percentage of subjects achieving treatment target of HbA1c less than 7.0% or less than or equal to 6.5% at Week 78 (end of treatment)
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 200 | 186
percentage (%) of subjects
  Treatment target HbA1c < 7% | 47 | 48
  Treatment target HbA1c =< 6.5% | 31 | 35

6. Secondary Outcome: Change in Body Weight at Week 26
Description: Change in body weight from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 231 | 229
kg | -3.24 (0.33) | -2.87 (0.33)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; ANCOVA model included treatment, country and previous treatment as fixed effects and baseline body weight as covariate. The objective was to demonstrate that treatment with liraglutide was different from treatment with exenatide. Thus the null hypothesis and its alternative were H0: µliraglutide = µexenatide against HA1:µliraglutide ≠ µexenatide where µliraglutide and µexenatide is the mean value of the body weight in the liraglutide arm and exenatide arm, respectively; Test type: Superiority or Other; p = 0.2235, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.38, 95% CI [-0.99 to 0.23]

7. Secondary Outcome: Change in Body Weight, Weeks 26-78
Description: Change in body weight from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group)
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 184
kg | -0.4 (3.24) | -0.7 (3.67)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; The analysis was made with a paired t test within the treatment group and 95% CIs for the difference between Weeks 26 and 78 were constructed. H0 was µ78 - µ26=0 against HA: µ78 - µ26 ≠ 0. A difference between the two means was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p = 0.0793, Paired t test; Mean = -0.4, 95% CI [-0.86 to 0.05], Standard Deviation 3.24
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; A paired t test was made within the group and 95% confidence intervals for the difference between Weeks 26 and 78 were constructed. H0 was µ78 - µ26 = 0 against HA: µ78 - µ26 ≠ 0. A difference between the two means (Week 26 and Week 78) was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p = 0.0075, Paired t test; Mean = -0.7, 95% CI [-1.26 to -0.20], Standard Deviation 3.67

8. Secondary Outcome: Change in Body Weight at Week 78
Description: Change in body weight from baseline (Week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group)
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 184
kg | -3.3 (4.63) | -3.2 (4.44)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; The analysis was made with a paired t test within the treatment group and 95% CIs for the difference between Weeks 0 and 78 were constructed. H0 was µ78- µ0=0 against HA: µ78 - µ0 ≠ 0. A difference between the two means was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -3.3, 95% CI [-3.90 to -2.61], Standard Deviation 4.63
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -3.2, 95% CI [-3.85 to -2.55], Standard Deviation 4.44

9. Secondary Outcome: Change in Fasting Plasma Glucose at Week 26
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 225 | 219
mmol/L | -1.61 (0.20) | -0.60 (0.20)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; ANCOVA model included treatment, country and previous treatment as fixed effects and baseline fasting plasma glucose as covariate. The objective was to demonstrate that treatment with liraglutide was different from treatment with exenatide. Thus the null hypothesis and its alternative were H0: µliraglutide = µexenatide against HA1:µliraglutide ≠ µexenatide where µliraglutide and µexenatide is the mean value of the fasting plasma glucose in the liraglutide and exenatide arm, respectively; Test type: Superiority or Other; p < 0.0001, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -1.01, 95% CI [-1.37 to -0.65]

10. Secondary Outcome: Change in Fasting Plasma Glucose, Weeks 26-78
Description: Change in fasting plasma glucose from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group)
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 197 | 182
mmol/L | 0.7 (1.84) | -0.1 (2.42)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; The analysis was made with a paired t test within the treatment group and 95% CIs for the difference between Weeks 26 and 78 were constructed. H0 was µ78- µ26=0 against HA: µ78 - µ26 ≠ 0. A difference between the two means was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = 0.7, 95% CI [0.48 to 1.00], Standard Deviation 1.84
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.4864, Paired t test; Mean = -0.1, 95% CI [-0.48 to 0.23], Standard Deviation 2.42

11. Secondary Outcome: Change in Fasting Plasma Glucose at Week 78
Description: Change in fasting plasma glucose from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group)
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 197 | 182
mmol/L | -1.3 (2.50) | -0.8 (2.76)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; The analysis was made with a paired t test within the treatment group and 95% CIs for the difference between Weeks 0 and 78 were constructed. H0 was µ78 - µ0=0 against HA: µ78 - µ0 ≠ 0. A difference between the two means was concluded when H0 was rejected at the 5% level; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -1.3, 95% CI [-1.62 to -0.92], Standard Deviation 2.50
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -0.8, 95% CI [-1.23 to -0.42], Standard Deviation 2.76

12. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Breakfast at Week 26
Description: Change in mean prandial increment of plasma glucose after breakfast from baseline (week 0) to 26 weeks (end of randomisation). Prandial increments of plasma glucose were calculated as the difference between glucose values measured before and after breakfast.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 207 | 196
mmol/L | -0.83 (0.28) | -2.16 (0.28)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; ANCOVA model included treatment, country and previous treatment as fixed effects and baseline value of the endpoint as covariate. The objective was to demonstrate that treatment with liraglutide was different from treatment with exenatide. Thus the null hypothesis and its alternative were H0: µliraglutide = µexenatide against HA1:µliraglutide ≠ µexenatide where µliraglutide and µexenatide is the mean value of the endpoint in the liraglutide arm and exenatide arm, respectively; Test type: Superiority or Other; p < .0001, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = 1.33, 95% CI [0.80 to 1.86]

13. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Lunch at Week 26
Description: Change in mean prandial increment of plasma glucose after lunch from baseline (week 0) to 26 weeks (end of randomisation). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after lunch.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 207 | 196
mmol/L | 0.06 (0.28) | 0.06 (0.28)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.9849, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = 0.01, 95% CI [-0.52 to 0.53]

14. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Dinner at Week 26
Description: Change in mean prandial increment of plasma glucose after dinner from baseline (week 0) to 26 weeks (end of randomisation). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after dinner.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 204 | 196
mmol/L | -1.10 (0.31) | -2.11 (0.31)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0005, ANCOVA — There were no multiplicity concerns; LS Mean = 1.01, 95% CI [0.44 to 1.57]

15. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Breakfast, Weeks 26-78
Description: Change in mean prandial increment of plasma glucose after breakfast from Week 26 (end of randomisation) to Week 78 (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after breakfast.
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 191 | 173
mmol/L | -0.22 (2.866) | 1.15 (3.253)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.2972, Paired t test; Mean = -0.22, 95% CI [-0.626 to 0.192], Standard Deviation 2.866
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = 1.15, 95% CI [0.660 to 1.637], Standard Deviation 3.253

16. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Lunch, Weeks 26-78
Description: Change in mean prandial increment of plasma glucose after lunch from Week 26 (end of randomisation) to Week 78 (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after a lunch.
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 191 | 173
mmol/L | 0.05 (3.307) | -0.09 (3.419)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.8396, Paired t test; Mean = 0.05, 95% CI [-0.424 to 0.521], Standard Deviation 3.307
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.7278, Paired t test; Mean = -0.09, 95% CI [-0.604 to 0.423], Standard Deviation 3.419

17. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Dinner, Weeks 26-78
Description: Change in mean prandial increment of plasma glucose after dinner from Week 26 (end of randomisation) to Week 78 (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after dinner.
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 190 | 172
mmol/L | 0.22 (3.053) | 1.07 (3.775)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.3271, Paired t test; Mean = 0.22, 95% CI [-0.219 to 0.654], Standard Deviation 3.053
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.0003, Paired t test; Mean = 1.07, 95% CI [0.497 to 1.634], Standard Deviation 3.775

18. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Breakfast at Week 78
Description: Change in mean prandial increment of plasma glucose after breakfast from baseline (week 0) to 78 weeks (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after breakfast.
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 192 | 167
mmol/L | -1.08 (3.662) | -0.99 (3.467)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -1.08, 95% CI [-1.605 to -0.562], Standard Deviation 3.662
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0003, Paired t test; Mean = -0.99, 95% CI [-1.517 to -0.458], Standard Deviation 3.467

19. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Lunch at Week 78
Description: Change in mean prandial increment of plasma glucose after lunch from baseline (week 0) to 78 weeks (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after lunch.
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 192 | 168
mmol/L | 0.26 (4.158) | -0.37 (3.838)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.3859, Paired t test; Mean = 0.26, 95% CI [-0.331 to 0.853], Standard Deviation 4.158
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2119, Paired t test; Mean = -0.37, 95% CI [-0.956 to 0.214], Standard Deviation 3.838

20. Secondary Outcome: Change in Mean Prandial Increment of Plasma Glucose After Dinner at Week 78
Description: Change in mean prandial increment of plasma glucose after dinner from baseline (week 0) to 78 weeks (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after dinner.
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 190 | 166
mmol/L | -0.35 (3.975) | -0.95 (3.230)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2290, Paired t test; Mean = -0.35, 95% CI [-0.917 to 0.2211], Standard Deviation 3.975
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0002, Paired t test; Mean = -0.95, 95% CI [-1.449 to -0.459], Standard Deviation 3.230

21. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Breakfast at Week 26
Description: Change in mean postprandial increment of plasma glucose after breakfast from baseline (week 0) to 26 weeks (end of randomisation). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after breakfast.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 207 | 197
mmol/L | -3.20 (0.31) | -3.93 (0.30)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0124, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = 0.73, 95% CI [0.16 to 1.31]

22. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Lunch at Week 26
Description: Change in mean postprandial increment of plasma glucose after lunch from baseline (week 0) to 26 weeks (end of randomisation). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after lunch.
Time Frame: week 0. week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 208 | 196
mmol/L | -2.74 (0.28) | -2.35 (0.28)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.1430, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.39, 95% CI [-0.91 to 0.13]

23. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Dinner at Week 26
Description: Change in mean postprandial increment of plasma glucose after dinner from baseline (week 0) to 26 weeks (end of randomisation). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after dinner.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 206 | 197
mmol/L | -3.05 (0.28) | -3.59 (0.27)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0380, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = 0.54, 95% CI [0.03 to 1.05]

24. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Breakfast, Weeks 26-78
Description: Change in mean postprandial increment of plasma glucose after breakfast from Week 26 (end of randomisation) to Week 78 (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after breakfast.
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 191 | 173
mmol/L | 0.06 (2.827) | 0.72 (3.270)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.7700, Paired t test; Mean = 0.06, 95% CI [-0.344 to 0.463], Standard Deviation 2.827
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0042, Paired t test; Mean = 0.72, 95% CI [0.230 to 1.212], Standard Deviation 3.270

25. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Lunch, Weeks 26-78
Description: Change in mean postprandial increment of plasma glucose after lunch from Week 26 (end of randomisation) to Week 78 (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after lunch.
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 191 | 173
mmol/L | 0.67 (3.041) | -0.09 (2.989)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.0026, Paired t test; Mean = 0.67, 95% CI [0.238 to 1.106], Standard Deviation 3.041
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6845, Paired t test; Mean = -0.09, 95% CI [-0.541 to 0.356], Standard Deviation 2.989

26. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Dinner, Weeks 26-78
Description: Change in mean postprandial increment of plasma glucose after dinner from Week 26 (end of randomisation) to Week 78 (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after dinner.
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 191 | 172
mmol/L | 0.32 (2.705) | 0.58 (3.114)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.1041, Paired t test; Mean = 0.32, 95% CI [-0.066 to 0.706], Standard Deviation 2.705
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0151, Paired t test; Mean = 0.58, 95% CI [0.114 to 1.052], Standard Deviation 3.114

27. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Breakfast at Week 78
Description: Change in mean postprandial increment of plasma glucose after breakfast from baseline (week 0) to 78 weeks (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after breakfast.
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 192 | 168
mmol/L | -3.31 (3.857) | -3.13 (3.560)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -3.31, 95% CI [-3.861 to -2.763], Standard Deviation 3.857
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -3.13, 95% CI [-3.673 to -2.589], Standard Deviation 3.560

28. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Lunch at Week 78
Description: Change in mean postprandial increment of plasma glucose after lunch from baseline (week 0) to 78 weeks (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after lunch.
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 192 | 168
mmol/L | -1.93 (3.703) | -2.17 (3.654)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -1.93, 95% CI [-2.457 to -1.403], Standard Deviation 3.703
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -2.17, 95% CI [-2.731 to -1.618], Standard Deviation 3.654

29. Secondary Outcome: Change in Mean Postprandial Increment of Plasma Glucose After Dinner at Week 78
Description: Change in mean postprandial increment of plasma glucose after dinner from baseline (week 0) to 78 weeks (end of treatment). Prandial increments of plasma glucose were calculated as the difference between plasma glucose values measured before and after dinner.
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 191 | 167
mmol/L | -2.21 (3.752) | -2.55 (3.625)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -2.21, 95% CI [-2.747 to -1.676], Standard Deviation 3.752
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -2.55, 95% CI [-3.104 to -1.997], Standard Deviation 3.625

30. Secondary Outcome: Change in Beta-cell Function at Week 26
Description: Change in Beta-cell function from baseline (week 0) to 26 weeks (end of randomisation). Beta-cell function was derived from fasting plasma glucose (FPG) and fasting insulin concentrations using the homeostasic model assessment (HOMA) method which uses the assumption that normal-weight normal subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
  Beta-cell function: HOMA-B (%) = 20∙fasting insulin[uU/mL] divided by (FPG mmol/L]-3.5).
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point (%point)
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 214 | 214
percentage point (%point) | 32.12 (6.75) | 2.74 (6.75)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = 29.37, 95% CI [16.81 to 41.93]

31. Secondary Outcome: Change in Beta-cell Function, Weeks 26-78
Description: Change in Beta-cell function from Week 26 (end of randomisation) to Week 78 (end of treatment). Beta-cell function was derived from fasting plasma glucose (FPG) and fasting insulin concentrations using the homeostasic model assessment (HOMA) method which uses the assumption that normal-weight normal subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
  Beta-cell function: HOMA-B (%) = 20∙fasting insulin[uU/mL] divided by (FPG mmol/L]-3.5).
Time Frame: week 26, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage point (%point)
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 179
percentage point (%point) | -18.18 (62.811) | 2.29 (52.997)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -18.18, 95% CI [-26.988 to -9.382], Standard Deviation 62.811
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5304, Paired t test; Mean = 2.49, 95% CI [-5.327 to 10.307], Standard Deviation 52.997

32. Secondary Outcome: Change in Beta-cell Function at Week 78
Description: Change in Beta-cell function from baseline (week 0) to 78 weeks (end of treatment). Beta-cell function was derived from fasting plasma glucose (FPG) and fasting insulin concentrations using the homeostasic model assessment (HOMA) method which uses the assumption that normal-weight normal subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
  Beta-cell function: HOMA-B (%) = 20∙fasting insulin[uU/mL] divided by (FPG mmol/L]-3.5).
Time Frame: week 0, week 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage point (%point)
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 189 | 176
percentage point (%point) | 24.86 (59.326) | 11.13 (87.145)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = 24.86, 95% CI [16.348 to 33.374], Standard Deviation 59.326
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0920, Paired t test; Mean = 11.13, 95% CI [-1.835 to 24.093], Standard Deviation 87.145

33. Secondary Outcome: Change in Total Cholesterol at Week 26
Description: Change in total cholesterol (TC) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 226 | 220
mmol/L | -0.20 (0.07) | -0.09 (0.07)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0946, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.11, 95% CI [-0.23 to 0.02]

34. Secondary Outcome: Change in Total Cholesterol, Weeks 26-78
Description: Change in total cholesterol (TC) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: Intention to Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects who entered the extension period and who had been exposed to at least one dose of the trial products.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 184
mmol/L | 0.11 (0.774) | 0.12 (0.804)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.0513, Paired t test; Mean = 0.11, 95% CI [-0.001 to 0.216], Standard Deviation 0.774
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.0513, Paired t test; Mean = 0.12, 95% CI [-0.001 to 0.233], Standard Deviation 0.804

35. Secondary Outcome: Change in Total Cholesterol at Week 78
Description: Change in total cholesterol (TC) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: Intention to Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects who entered the extension period and who had been exposed to at least one dose of the study products.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 183
mmol/L | -0.07 (0.859) | 0.09 (0.890)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2764, Paired t test; Mean = -0.07, 95% CI [-0.187 to 0.054], Standard Deviation 0.859
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.1911, Paired t test; Mean = 0.09, 95% CI [-0.043 to 0.216], Standard Deviation 0.890

36. Secondary Outcome: Change in Low-density Lipoprotein-cholesterol at Week 26
Description: Change in Low-density Lipoprotein-cholesterol (LDL-C) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 219 | 215
mmol/L | -0.44 (0.06) | -0.40 (0.06)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.4412, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.04, 95% CI [-0.15 to 0.06]

37. Secondary Outcome: Change in Low-density Lipoprotein-cholesterol, Weeks 26-78
Description: Change in low-density lipoprotein-cholesterol (LDL-C) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 180
mmol/L | 0.03 (0.606) | 0.08 (0.720)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.4746, Paired t test; Mean = 0.03, 95% CI [-0.054 to 0.115], Standard Deviation 0.606
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1281, Paired t test; Mean = 0.08, 95% CI [-0.024 to 0.188], Standard Deviation 0.720

38. Secondary Outcome: Change in Low-density Lipoprotein-cholesterol at Week 78
Description: Change in Low-density Lipoprotein-cholesterol (LDL-C) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 183 | 176
mmol/L | -0.30 (0.604) | -0.21 (0.647)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -0.30, 95% CI [-0.390 to -0.214], Standard Deviation 0.604
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -0.21, 95% CI [-0.303 to -0.110], Standard Deviation 0.647

39. Secondary Outcome: Change in Very Low-density Lipoprotein-cholesterol at Week 26
Description: Change in very low-density lipoprotein-cholesterol (VLDL-C) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 216 | 212
mmol/L | 0.20 (0.04) | 0.27 (0.04)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0277, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.07, 95% CI [-0.13 to -0.01]

40. Secondary Outcome: Change in Very Low-density Lipoprotein-cholesterol, Weeks 26-78
Description: Change in Very Low-density Lipoprotein-cholesterol (VLDL-C) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 180
mmol/L | 0.06 (0.290) | 0.03 (0.307)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.0030, Paired t test; Mean = 0.06, 95% CI [0.021 to 0.102], Standard Deviation 0.290
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1452, Paired t test; Mean = 0.03, 95% CI [-0.012 to 0.079], Standard Deviation 0.307

41. Secondary Outcome: Change in Very Low-density Lipoprotein-cholesterol at Week 78
Description: Change in Very Low-density Lipoprotein-cholesterol (VLDL-C) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 173 | 168
mmol/L | 0.27 (0.306) | 0.31 (0.346)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = 0.27, 95% CI [0.223 to 0.315], Standard Deviation 0.306
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = 0.31, 95% CI [0.259 to 0.364], Standard Deviation 0.346

42. Secondary Outcome: Change in High-density Lipoprotein-cholesterol at Week 26
Description: Change in High-density Lipoprotein-cholesterol (HDL-C) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 226 | 220
mmol/L | -0.04 (0.02) | -0.05 (0.02)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.5105, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = 0.01, 95% CI [-0.02 to 0.04]

43. Secondary Outcome: Change in High-density Lipoprotein-cholesterol, Weeks 26-78
Description: Change in High-density Lipoprotein-cholesterol (HDL-C) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 119 | 180
mmol/L | -0.01 (0.150) | 0.00 (0.141)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.2220, Paired t test; Mean = -0.01, 95% CI [-0.034 to 0.008], Standard Deviation 0.150
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7923, Paired t test; Mean = 0.00, 95% CI [-0.018 to 0.024], Standard Deviation 0.141

44. Secondary Outcome: Change in High-density Lipoprotein-cholesterol at Week 78
Description: Change in High-density Lipoprotein-cholesterol (HDL-C) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 183 | 176
mmol/L | -0.03 (0.159) | -0.02 (0.165)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0254, Paired t test; Mean = -0.03, 95% CI [-0.050 to -0.003], Standard Deviation 0.159
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2244, Paired t test; Mean = -0.02, 95% CI [-0.040 to 0.009], Standard Deviation 0.165

45. Secondary Outcome: Change in Triglyceride at Week 26
Description: Change in triglyceride (TG) from from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 225 | 220
mmol/L | -0.41 (0.10) | -0.23 (0.10)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0485, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.18, 95% CI [-0.37 to -0.00]

46. Secondary Outcome: Change in Triglyceride, Weeks 26-78
Description: Change in Triglyceride (TG) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 184
mmol/L | 0.1 (0.82) | -0.0 (0.96)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.1161, Paired t test; Mean = 0.1, 95% CI [-0.02 to 0.21], Standard Deviation 0.82
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7888, Paired t test; Mean = -0.0, 95% CI [-0.16 to 0.12], Standard Deviation 0.96

47. Secondary Outcome: Change in Triglyceride at Week 78
Description: Change in triglyceride (TG) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 183
mmol/L | -0.3 (1.07) | -0.1 (1.47)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0003, Paired t test; Mean = -0.3, 95% CI [-0.43 to -0.13], Standard Deviation 1.07
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2078, Paired t test; Mean = -0.1, 95% CI [-0.35 to 0.08], Standard Deviation 1.47

48. Secondary Outcome: Change in Free Fatty Acid at Week 26
Description: Change in Free Fatty Acid (FFA) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 220 | 222
mmol/L | -0.17 (0.02) | -0.10 (0.02)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0014, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.07, 95% CI [-0.11 to -0.03]

49. Secondary Outcome: Change in Free Fatty Acid, Weeks 26-78
Description: Change in Free Fatty Acid (FFA) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 182
mmol/L | 0.06 (0.269) | 0.01 (0.272)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.0018, Paired t test; Mean = 0.06, 95% CI [0.023 to 0.098], Standard Deviation 0.269
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5499, Paired t test; Mean = 0.01, 95% CI [-0.028 to 0.052], Standard Deviation 0.272

50. Secondary Outcome: Change in Free Fatty Acid at Week 78
Description: Change in Free Fatty Acid (FFA) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 195 | 182
mmol/L | -0.10 (0.273) | -0.07 (0.302)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -0.10, 95% CI [-0.140 to -0.062], Standard Deviation 0.273
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0012, Paired t test; Mean = -0.07, 95% CI [-0.118 to -0.030], Standard Deviation 0.302

51. Secondary Outcome: Change in Apolipoprotein B at Week 26
Description: Change in apolipoprotein B (ApoB) from baseline (week 0) to 26 weeks (end of randomisation)
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 226 | 222
g/L | -0.06 (0.02) | -0.03 (0.02)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide vs Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.1119, ANCOVA — There were no multiplicity concerns; Estimated treatment difference, LS Mean = -0.02, 95% CI [-0.05 to 0.01]

52. Secondary Outcome: Change in Apolipoprotein B, Weeks 26-78
Description: Change in apolipoprotein B (ApoB) from Week 26 (end of randomisation) to Week 78 (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 26, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 199 | 184
g/L | -0.02 (0.168) | -0.03 (0.189)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.1342, Paired t test; Mean = -0.02, 95% CI [-0.041 to 0.006], Standard Deviation 0.168
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0344, Paired t test; Mean = -0.03, 95% CI [-0.057 to -0.002], Standard Deviation 0.189

53. Secondary Outcome: Change in Apolipoprotein B at Week 78
Description: Change in apolipoprotein B (ApoB) from baseline (week 0) to 78 weeks (end of treatment) within each treatment group (the liraglutide -> liraglutide group and the exenatide -> liraglutide group).
Time Frame: week 0, week 78
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 198 | 184
g/L | -0.08 (0.176) | -0.07 (0.192)
Statistical Analysis 1: Comparison: Liraglutide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -0.08, 95% CI [-0.105 to -0.056], Standard Deviation 0.176
Statistical Analysis 2: Comparison: Exenatide -> Liraglutide -> Liraglutide; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t test; Mean = -0.07, 95% CI [-0.094 to -0.038], Standard Deviation 0.192

54. Secondary Outcome: Hypoglycaemic Episodes at Week 26
Description: Total number of hypoglycaemic episodes occurring after baseline (week 0) and until week 26 (end of randomisation). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: weeks 0-26
Population: The safety analysis set is all subjects who had been exposed to at least one dose of the study products.
Measure: Number; unit: episodes
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 235 | 232
episodes
  Major | 0 | 2
  Minor | 208 | 264
  Symptoms only | 79 | 93

55. Secondary Outcome: Hypoglyceamic Episodes, Weeks 26-78
Description: Total number of hypoglycaemic episodes occurring after end of randomisation (week 26) and until week 78 (end of treatment). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: weeks 26-78
Population: The safety analysis set is all subjects who had been exposed to at least one dose of the study products.
Measure: Number; unit: episodes
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Number analyzed (Participants) | 202 | 187
episodes
  Major | 1 | 0
  Minor | 140 | 172
  Symptoms only | 37 | 32

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time span of 78 weeks.
Description: The safety analysis set included all subjects who had been exposed to at least one dose of the study products.
Arm/Group | Liraglutide -> Liraglutide -> Liraglutide | Exenatide -> Liraglutide -> Liraglutide
Serious Adverse Events (participants affected / at risk) | 23/235 | 23/232
Other Adverse Events (participants affected / at risk) | 162/235 | 167/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide -> Liraglutide -> Liraglutide (N=235) | Exenatide -> Liraglutide -> Liraglutide (N=232)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Blood product transfusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide -> Liraglutide -> Liraglutide (N=235) | Exenatide -> Liraglutide -> Liraglutide (N=232)
Anorexia (Metabolism and nutrition disorders) | 10 (10) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (30) | 12 (13)
Bronchitis (Infections and infestations) | 15 (18) | 20 (22)
Constipation (Gastrointestinal disorders) | 18 (18) | 10 (13)
Diarrhoea (Gastrointestinal disorders) | 35 (47) | 37 (50)
Dizziness (Nervous system disorders) | 14 (16) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 25 (35) | 14 (17)
Headache (Nervous system disorders) | 29 (38) | 28 (40)
Hypertension (Vascular disorders) | 10 (10) | 12 (12)
Influenza (Infections and infestations) | 13 (14) | 11 (11)
Nasopharyngitis (Infections and infestations) | 43 (59) | 42 (71)
Nausea (Gastrointestinal disorders) | 64 (87) | 68 (92)
Sinusitis (Infections and infestations) | 12 (14) | 9 (13)
Upper respiratory tract infection (Infections and infestations) | 26 (33) | 28 (30)
Vomiting (Gastrointestinal disorders) | 19 (20) | 26 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.